CLINICAL TRIAL: NCT00768573
Title: A Single-Blind Study In Healthy Adult Volunteers To Investigate The Palatability Of Different Oral Suspension Formulations Of Revatio®
Brief Title: Taste Test of a New Formulation of Sildenafil (Revatio)
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481257
Record Dates: First submitted 2008-09-04; First posted 2008-10-08 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: None Volunteer
Keywords: taste test
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1. Taste test
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: sildenafil — Oral suspension of sildenafil.

SUMMARY:
taste of formulation

DETAILED DESCRIPTION:
taste test None

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* History of hypersensitivity to test compounds or excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
palatability (aroma, flavour texture and mouth feel) | Duration of study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Cambridge, Massachusetts, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481257&StudyName=Taste%20test%20of%20a%20new%20formulation%20of%20sildenafil%20%28revatio%29.